CLINICAL TRIAL: NCT04259619
Title: Low-Level-Lasertherapie (LLLT) Bei Schmerzhaften, Wunden Mamillen Stillender Frauen
Brief Title: Low-Level Laser Therapy (LLLT) Treatment for Breast-Feeding Women With Painful Nipple Lesions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-01374
Record Dates: First submitted 2020-02-05; First posted 2020-02-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Nipple Lesions
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: prospective, randomized double-blinded study
Who Masked: Participant, Care Provider, Investigator
Masking Description: The low-level laser and the placebo-laser cannot be differentiated visually. The lasers are marked with the names "Geraet1" and "Geraet2". The therapy is carried out identical in the way of application, duration and preventive measures. After the participant is randomized, the study nurse hands out the corresponding laser for the therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Level Laser Therapy (Experimental): During 2-3 days this group receives three low-level laser therapy (LLLT) treatments with the Soft Power Laser carried out by a specially trained breastfeeding consultant.
  Interventions: Device: Low-Level Laser Therapy
- Placebo Therapy (Placebo Comparator): During 2-3 days this group receives three placebo treatments with an identically looking laser, which in contrast submits only red colored light. The therapy is also carried out by a specially trained breastfeeding consultant.
  Interventions: Device: Placebo Therapy

INTERVENTIONS:
Device: Low-Level Laser Therapy — The low-level laser emits monochromatic, coherent, bundled laser light. In each therapy a energy dose of 2-4 Joul (J) / centimeter (cm)^2 is applied over a duration of about 30 seconds using level 1 (20 percent of maximum output) of the 350 milliwatt (mW) device.
  Arms: Low-Level Laser Therapy
Device: Placebo Therapy — The intervention is conducted identically to the low-level laser therapy but the placebo laser that is used emits only red light that is polychromatic, leading to a reduction in energy being emitted and therewith to no or a smaller effect.
  Arms: Placebo Therapy

SUMMARY:
Around 30 to 90 percent of all breastfeeding women suffer from painful and sore nipple lesions. Reasons for these lesions are still not completely clarified. Nevertheless, irrespective of the underlying cause, these painful nipple lesions lead to an early stop of breastfeeding, which has negative consequences for the infant as well as for the mother. Even if the painful nipple lesions do not lead to a weaning of the baby, they cause an increased psychological distress for the mother and therefore may negatively influence the mother-child relationship.

Since breastfeeding is the natural and best possible type of nutrition for healthy, full term babies problems causing an early stop of breastfeeding should be addressed.

The low-level laser therapy (LLLT) represents a simple and low risk treatment to change (reduce) pain and accelerate wound healing. It is supposed to improve tissue organization and should have a positive anti-inflammatory and immune modulating effect. Therefore, this therapy is more and more frequently used to also treat painful nipple lesions, although hardly any studies have been conducted. Furthermore, in women with too little mother milk, the LLLT seems to increase the milk production.

The aim of this study is to investigate the positive effects of LLLT on painful and sore nipple lesions. This would justify a LLLT for women with painful nipple lesions on a wider scale, with the overall goal to reduce early stopping of breastfeeding and therefore having a positive impact on both, the child's health as well as the mother's wellbeing.

DETAILED DESCRIPTION:
This study is conducted at the department of obstetrics of the University hospital of Zurich. 194 breastfeeding or expressing participants with sore and painful nipple lesions who fulfill the inclusion criteria are included in this study. If the participant meets any exclusion criteria she is excluded from this study. After being enrolled in the study, the participant is randomized to get either 3 low-level laser therapy (LLLT) treatments or 3 placebo treatments within 1 to 3 days.

Women having signed the declaration of consent and fulfill all inclusion criteria are then examined by a breastfeeding consultant. During this examination nipple lesions are classified into four different stages, causes for the lesions are evaluated and the nipple form is recorded. A swab of the milk is taken to rule out a pathogenetic colonization with germs. Then a blood sample is collected to analyze inflammatory parameters (C-reactive protein (CRP), leucocyte (Lc)), inflammation modulators (interleukin 6 (IL-6), tumor necrosis factor alpha (TNF-α)) and the lactating hormone (prolactin). The taking of blood is repeated at the end of the third therapy. In the beginning and at the end of the last treatment, nipple lesions are classified and photographically documented. Specific instructions regarding the correct positioning and removal of the baby at the breast as well as breastfeeding positions are given to the women before starting the treatment. Women then breastfeed their baby once before and once after the entire therapy. Two hours after breastfeeding, the amount of milk is being measured after 15 minutes of pumping. Additionally, the sensation of pain is evaluated on the basis of a visual analog scale (VAS) from 1-10 and the satisfaction of the treatment is recorded before and after every single treatment. At the end of the last therapy, a final examination is conducted.

For the statistical analysis of the primary and secondary endpoints a proportional odds model is used.

ELIGIBILITY:
Inclusion Criteria:

* signed written informed consent form
* breast-feeding or pumping participant with painful nipple lesions
* 18 years or older

Exclusion Criteria:

* contraindication for the class of medical device used or intervention being performed e.g.

known hypersensitivity or allergy against the medical device or class of medical device

* missing willingness to take part in the study
* hepatitis B or C positive
* human immunodeficiency virus (HIV) positive
* intake of immunosuppressive drugs
* epilepsy
* dark or tattooed skin
* lacking German or English skills
* mamma carcinoma in past medical history
* severe infection (C-reactive protein (CRP) >200mg/l; leucocytes >20000/ul)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2026-02-01 (Actual); Study Completion 2026-02-01 (Actual)

PRIMARY OUTCOMES:
Pain Reduction: visual pain scale from 1 (no pain) to 10 (worst pain) | though individual study completion, an average of 3 days
  The primary goal is to evaluate the pain change with the help of a visual pain scale form 1 to 10 (0 = no pain; 10 = worst pain).

SECONDARY OUTCOMES:
Wound Healing | though individual study completion, an average of 3 days
  One secondary goal is to evaluate the effect of the low-level laser therapy (LLLT) on wound healing. For this evaluation the nipple lesions are staged from 1-4 and photo documented and inflammatory markers (C reactive protein (CRP) and leucocytes (Lc)) and modulators (interleukin 6 (IL6) and tumor necrosis factor alpha (TNF-a) are analyzed in the blood.
Milk Production | though individual study completion, an average of 3 days
  Another secondary goal is to evaluate the effect of the low-level laser therapy (LLLT) on milk production. This is done through measuring the milk production after 15 minutes pumping of both breasts and analyzing the prolactin in the blood.
Satisfaction with the low-level laser therapy (LLLT): visual analogue scale from 1 (low satisfaction) to 10 (highest satisfaction) | though individual study completion, an average of 3 days
  An additional secondary goal is to evaluate the participants' degree of satisfaction with the LLLT. This is accomplished with the help of a visual analogue scaled.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Ochsenbein-Kölble, Prof.Dr.med., Principal Investigator — leading physician
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland